CLINICAL TRIAL: NCT06466590
Title: Reliability and Validity of the French Version of the Virtual Reality Sickness Questionnaire
Acronym: VRSQ-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A02468-37
Record Dates: First submitted 2024-06-07; First posted 2024-06-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Virtual Reality Cyber Sickness
Keywords: virtual reality; cyber sickness; assessment

STUDY DESIGN:
Intervention Model Description: All participants will perform 4 exercises in virtual reality with HMD (Head Mounted Display). Then, they will use the VRSQ-F instrument under study on 2 times separated by 15 minutes. The primary objective is to assess the reliability and validity of this instrument through repeated measures and comparison to SSQ
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Group (Experimental): Participants will be asked to use the measurement instrument VRSQ-F on two separate occasions under identical conditions to assess its test-retest reliability and asked to use the SSQ for validity. Each session will involve completing the measurement protocol as specified.
  Interventions: Diagnostic Test: Use of Measurement Instrument

INTERVENTIONS:
Diagnostic Test: Use of Measurement Instrument — Participants will complete the measurement procedure twice, with sessions scheduled one week apart, using the same instrument under standardized conditions. The results from both sessions will be compared to assess the instrument's consistency and accuracy

SUMMARY:
This is a multicenter, controlled, non-randomized interventional clinical study, with minimal risks and constraints, aimed at verifying the reliability of the French version of the VRSQ questionnaire (VRSQ-F) and the validity of the VRSQ-F score by comparing it with the SSQ score.

ELIGIBILITY:
Inclusion Criteria:

For Healthy people :

* Men or women aged 18 to 65
* Person affiliated to a social security scheme
* Healthy person with no particular medical condition
* Having given their consent to participate in the research

For patients :

* Men or women aged 18 to 65
* Persons affiliated to a social security scheme
* People undergoing regular rehabilitation, walking or in a wheelchair, who can use a virtual reality solution as part of their care.
* Having given their consent to take part in the research

Exclusion Criteria:

* Vestibular and cardiac pathologies, and major visual disorders not compatible with virtual reality rehabilitation
* Cognitive and language disorders
* Persons under legal protection
* Pregnant women
* MSSQ greater than 15
* People suffering from photosensitive epilepsy
* Persons under the influence of medication that may impair drugs or alcohol
* Participant with an implanted medical device that may be affected by radio waves emitted by compatible third-party equipment (e.g. : Pacemaker)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Check the validity of the VRSQ-F score by comparing it with the SSQ score | Immediately after exercises
  Criteria validity between SSQ and VRSQ-F. SSQ questionnaire with 16 questions scoring from 0 to 48 VRSQ-F questionnaire with 9 questions from 0 to 27
Reliability of VRSQ-F (Virtual Reality Sickness Questionnaire) using the intraclass correlation coefficient between measurements immediately after VR exercises and 15 min after and Cronbach coefficient of the VRSQ-F questionnaire | Immediately after exercises
  Reliability of VRSQ-F (Virtual Reality Sickness Questionnaire) using the intraclass correlation coefficient between measurements immediately after VR exercises and 15 min after and Cronbach coefficient of the VRSQ-F questionnaire

SECONDARY OUTCOMES:
Calculate the minimum detectable change in the questionnaire | Immediately after exercises
  Clinimetric quality: Calculation of the standard error of measurement SEM and the minimum detectable change MDC

CONTACTS AND LOCATIONS:
Overall Officials: Emilie LEBLONG, Principal Investigator — Pôle Saint Hélier
Locations (3):
- France (3):
  - Centre de Rééducation Fonctionnelle Neurologique PROPARA, Montpellier
  - Pôle Saint-Hélier, Rennes
  - Fondation Ildys, Roscoff